CLINICAL TRIAL: NCT04099329
Title: One Team: Changing the Culture of Youth Sport With Pregame Safety Huddles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Georgia Southern University (Other); University of Oregon (Other); Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Principal Investigator, Sara PD Chrisman, MD MPH, Associate Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00000972
Record Dates: First submitted 2019-08-07; First posted 2019-09-23 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Concussion, Brain
Keywords: Soccer; Football; Injury; Prevention; Concussion; Education; Huddles; Primary prevention; Secondary prevention; Behavioral intervention
MeSH Terms: conditions — Brain Concussion; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Leagues were randomized to intervention or control
Who Masked: Investigator
Masking Description: Data masked for analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-game Safety Huddles (Experimental): Pre-game safety huddles will occur before each game and athletes and coaches will be surveyed.
  Interventions: Behavioral: Pre-game Safety Huddles
- Control (No Intervention): No intervention will be delivered by athletes and coaches will be surveyed.

INTERVENTIONS:
Behavioral: Pre-game Safety Huddles — Coaches will be trained to lead Pre-game Safety Huddles by the RA with the study using a multi-media tool we have developed. Huddles will be brief (1-2 minutes) and will primarily focused on 1) encouraging concussion reporting and 2) encouraging good sportsmanship
  Arms: Pre-game Safety Huddles

SUMMARY:
Randomized controlled trial of a behavioral intervention (Pre-Game Safety Huddles) designed to study the impact of huddles on concussion safety in youth sport, primarily regarding intention to report concussive symptoms.

DETAILED DESCRIPTION:
More than 1 million youth sustain a sport-related concussion (SRC) each year. The middle school age range is particularly concerning because it is a time when children have both a unique susceptibility to brain injury and high participation rates in organized sports with concussion risk, such as soccer and football. There are two avenues to decrease concussion risk: (1) minimizing the number and force of collisions to decrease concussion incidence (primary prevention) and (2) improving concussion identification to decrease morbidity (secondary prevention). The goal of this study is to utilize Pre-Game Safety Huddles to discuss sportsmanship (primary prevention) and concussion reporting (secondary prevention) with a goal of improving concussion safety.

To assess the efficacy of Pre-Game Safety Huddles as a tool for injury prevention, we will conduct a Randomized controlled trial with youth sport teams. We will recruit leagues in the Seattle area (girls' soccer, boys' soccer and football) and randomize them to either intervention or control. Coaches in the intervention group will then be trained to lead Pre-Game Safety Huddles before each game over the course of the season (9-12 weeks). Youth and coaches will be surveyed at three time points and data will be analyzed to determine impact of the intervention on two outcomes: 1) expectations regarding reporting concussive symptoms (CR-E) and 2) expectations regarding engaging in potentially injurious play (IP-E).

ELIGIBILITY:
Inclusion Criteria:

* Participating on a team in one of the recruited leagues and willing to complete surveys

Exclusion Criteria:

* Not willing to complete surveys

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2019-08-24 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change, Expectations regarding concussion reporting (CR-E) | Baseline, 4-6 weeks, 9-12 weeks
  Self-report survey of Athlete expectations regarding reporting concussive symptoms

SECONDARY OUTCOMES:
Change, Expectations of engaging in potentially injurious play (IP-E) | Baseline, 4-6 weeks, 9-12 weeks
  Self-report survey of Athlete rating of expectations of engaging in potentially risky sport behavior
Change, Perceived coach, parent and peer norms regarding concussion reporting (PN-PWCS) | Baseline, 4-6 weeks, 9-12 weeks
  Self-report survey, Athlete perception of norms regarding concussion reporting
Change in Perceived coach (TN-C), parent (TN-P) and peer norms (TN-T) regarding sportsmanship | Baseline, 4-6 weeks, 9-12 weeks
  Self-report survey, Athlete perception of norms regarding sportsmanship
Change, Youth sport values (YSV) | Baseline, 4-6 weeks, 9-12 weeks
  Self-report survey, Athlete values regarding sport participation
Self-report of concussion diagnosis | 9-12 weeks
  Athlete report of concussion diagnosis during the season
Change, Expectations regarding reporting teammate concussion (bystander reporting) (E-BR) | Baseline, 4-6 weeks, 9-12 weeks
  Self-report survey, Athlete intention to report teammate concussive symptoms
Change, Prosocial and Antisocial Behavior in Sport Scale (PABSS) | Baseline, 4-6 weeks, 9-12 weeks
  Self-report survey, Standardized measure of sportsmanship
Performed behavior, concussion reporting (PB--CR) | 9-12 weeks
  Self-report survey, Athlete concussion symptoms following potential concussion during season
Acceptability of Intervention Measure (AIM-2) and Feasibility of Intervention Measure (AIM-2, FIM-2) | 9-12 weeks
  Self-report survey, Standardized measures of acceptability and feasibility

CONTACTS AND LOCATIONS:
Locations (1):
- Sara P Chrisman, Seattle, Washington, United States

REFERENCES:
- [Derived] Kroshus E, Chrisman SPD, Glang A, Hunt T, Hays R, Lowry S, Peterson A, Garrett K, Ramshaw D, Hafferty K, Kinney E, Manzueta M, Steiner MK, Bollinger BJ, Chiampas G, Rivara FP. Concussion education for youth athletes using Pre-Game Safety Huddles: a cluster-randomised controlled trial. Inj Prev. 2023 Feb;29(1):22-28. doi: 10.1136/ip-2022-044665. Epub 2022 Sep 16. PMID 36113984

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT04099329/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT04099329/ICF_001.pdf